CLINICAL TRIAL: NCT05883904
Title: Observational Study Protocol REALFed - Real World Evidence of Fedratinib Effectiveness in Myelofibrosis
Brief Title: Real World Evidence of Fedratinib Effectiveness in MF
Acronym: REALFed
Status: Recruiting | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: MPN0123
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Primary Myelofibrosis; Post-polycythemia Vera Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — fedratinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Fedratinib — Fedratinib administered after AIFA reimbusement approval

SUMMARY:
This is a multicenter prospective and retrospective observational clinical study in patients with primary or post polycythemia vera or post essential thrombocythemia myelofibrosis to test the efficacy of fedratinib in the rea world. Participants will be managed according to the clinical practice of the participating Center. All Centers will be Italian Hematology Units belonging to the GIMEMA Organization in Italy.

DETAILED DESCRIPTION:
This is a multicenter prospective and retrospective observational clinical study with the aim of assessing the efficacy of fedratinib upon AIFA approval in patients with primary myelofibrosis or post polycythemia vera or post essential thrombocythemia myelofibrosis. Patients must meet current diagnostic criteria of MF, according to the WHO (World Health Organization) classification version 5th or the ICC (International Consensus Conference) either published in 2022 or post- polycythemia vera and post-essential thrombocythemia myelofibrosis (according to the ICC classification 2022). Patients enter the study at diagnosis or already in follow-up, at any stage of disease, except if transformed to blast phase. Patients who received fedratinib after June 2022 (time of AIFA reimbursement in Italy) will be enrolled and will be included both those ruxolitinib-naïve and ruxolitinib-exposed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Patients diagnosed with primary myelofibrosis [according to the WHO (World Health Organization) classification version 5th or the ICC (International Consensus Conference) either published in 2022 or post-polycythemia vera and post-essential thrombocythemia myelofibrosis (according to the ICC classification 2022)].
* Patients who met the reimbursement criteria for fedratinib, in accordance with the AIFA (Agenzia Italiana del Farmaco) after June 2022.
* Patients eligible or not for stem cell transplant (SCT) or patients already undergoing SCT.
* Patients on non-JAKi cytoreductive treatment.
* Patients with palpable splenomegaly at baseline of fedratinib treatment.
* Informed consent signed, if applicable.

Exclusion Criteria:

* Diagnosis of MPN, unclassifiable, myelodysplastic/myeloproliferative neoplasms, myelodysplastic syndromes, essential thrombocythemia, polycythemia vera.
* Blast phase of MF.
* Patients with platelets <50 x10^9/L at baseline of fedratinib treatment.
* Patients ruxolitinib-exposed for other diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by MF, according to the WHO classification version 5th or the ICC ) or post- polycythemia vera and post-essential thrombocythemia myelofibrosis according to the ICC who received fedratinib after June 2022 (time of AIFA reimbursement in Italy) will be enrolled and will be included both those ruxolitinib-naïve and ruxolitinib-exposed.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Splenic response | 6 months
  Splenic response is defined as 50% palpatory reduction.

CONTACTS AND LOCATIONS:
Locations (1):
- Ematologia FONDAZIONE IRCCS CA' GRANDA, OSPEDALE MAGGIORE POLICLINICO, Milan, Italy